CLINICAL TRIAL: NCT03876821
Title: Collect of Cord Blood From Subjects at Risk for Sickle Cell Disease, for the Purpose of Laboratory Research
Acronym: DREPACORD
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: C18-31
Record Dates: First submitted 2019-02-27; First posted 2019-03-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-05

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from cord blood cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study consists in collecting umbilical cord blood cells from newborns at risk of sickle cell disease, to perform laboratory experiments aiming to characterize the cells with HbS/HbS mutation, to develop methods to prepare, to gene-modify and to preserve these cells.

DETAILED DESCRIPTION:
Pregnant individuals carrying at least one HbS allele will be included in the study to collect the umbilical cord blood of the child at birth. Collected cells will be used anonymously for genetic and bioexperimental laboratory research, aiming to develop autologous gene therapy for sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, giving birth at CHSF and consenting to the collect and study of placental blood after delivery
* Age 18 to 45 years
* Biological testing of the participant includes hemoglobin electrophoresis and shows at least one HbS allele

Exclusion Criteria:

* Lack of written consent
* Minors (not 18 years old) or under guardianship
* Diseases : HIV, Hepatitis B, Hepatitis C or HTLV (Human T Leukemia Virus).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Giving birth
Study Population: The study includes pregnant women, aged 18-45 years of age, carrying at least one HbS allele, and who are followed and giving birth at the maternity unit of the Centre Hospitalier Sud Francilien in Evry, France.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Number of samples with HbS/HbS genotype | 3 years
  Measured by DNA sequencing

SECONDARY OUTCOMES:
Number of samples with bio-experimental data | 4 years
  Consisting of cellular characterization, transduction and cell processing data

CONTACTS AND LOCATIONS:
Overall Officials: Luc Rigonnot, MD, Principal Investigator — CHSF; Anne Galy, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- CHSF, Corbeil-Essonnes, France

REFERENCES:
- [Result] Mormin M, Rigonnot L, Chalumeau A, Miccio A, Fournier C, Pajanissamy S, Dewannieux M, Galy A. Cyclosporin H Improves the Transduction of CD34+ Cells with an Anti-Sickling Globin Vector, a Possible Therapeutic Approach for Sickle Cell Disease. Hum Gene Ther. 2024 Nov;35(21-22):896-903. doi: 10.1089/hum.2024.098. Epub 2024 Nov 6. PMID 39504955